CLINICAL TRIAL: NCT00195338
Title: A Post-Marketing Surveillance Looking At Safety And Adherence To Treatment Of Enbrel In Adults With Active Rheumatoid Arthritis In Luxemburg
Brief Title: Study Evaluating Enbrel In Adults With Active Rheumatoid Arthritis In Luxemburg
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: Innovex, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 0881-101343
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2012-01-23 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2011-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: This is an open label, observational study.This is a post-marketing surveillance study in rheumatology practice patients in Luxemburg.Rheumatologists will be asked to document safety and adherence to therapy of Enbrel when given to adults with active rheumatoid arthritis.All patients initiated with Enbrel will be observed.
  Interventions: Drug: etanercept

INTERVENTIONS:
Drug: etanercept

SUMMARY:
The purpose of the study is to determine the long term safety of Enbrel in adults with active rheumatoid arthritis in Luxemburg. This is a post-marketing surveillance study in rheumatology practice patients. All patients initiated with Enbrel will be observed from the start of the study in Feb 2003 for a period of at least 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Have moderate to severe active rheumatoid arthritis
* Be aged of 17 years or more
* Have inadequate response to DMards
* Give written informed consent
* Physician decides to prescribe Enbrel

Exclusion Criteria:

n/a

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be included after the physician decided to prescribe Enbrel.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2004-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Luxembourg, Luxembourg

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881-101343&StudyName=Study%20Evaluating%20Enbrel%20In%20Adults%20With%20Active%20Rheumatoid%20Arthritis%20In%20Luxemburg

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept: Etanercept (Enbrel) injection administered subcutaneously (s.c.) as per scientific leaflet specifications.
Period: Overall Study
Arm/Group | Etanercept
Started | 25
Completed | 13
Not Completed | 12
Not completed — Lost to Follow-up | 2
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 1
Not completed — Early closure of the site | 4

BASELINE CHARACTERISTICS:
Arm/Group | Etanercept
Number analyzed (Participants) | 25
Age Continuous [Mean (Standard Deviation); unit: years] | 50.20 (13.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Any untoward medical occurrence in a participant who received study treatment was considered an AE without regard to possibility of causal relationship. An AE resulting in any of the following outcomes, or deemed to be significant for any other reason, was considered to be a SAE: death; initial or prolonged inpatient hospitalization; a life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline up to Month 66
Population: Full analysis set (FAS) included all recruited participants who were either initiated or were already receiving etanercept.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 25
percentage of participants
  AEs | 56
  SAEs | 24

2. Secondary Outcome: Percentage of Participants With Completion of Study Treatment
Time Frame: Month 12 through Month 72
Population: FAS included all recruited participants who were either initiated or were already receiving etanercept.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 25
percentage of participants
  12 to 18 months | 100
  Greater than 18 months to 24 months | 100
  Greater than 24 months to 30 months | 92
  Greater than 30 months to 36 months | 80
  Greater than 36 months to 42 months | 80
  Greater than 42 months to 48 months | 80
  Greater than 48 months to 54 months | 68
  Greater than 54 months to 60 months | 52
  Greater than 60 months to 66 months | 28
  Greater than 66 months to 72 months | 12
  Greater than 72 months | 12

3. Secondary Outcome: Change From Baseline in Number of Joints With Active Synovitis at Months 6, 12, 18, 30, 42, 54 and 66
Description: Synovitis was defined as the inflammation of a synovial (joint-lining) membrane, usually painful, particularly on motion, and characterized by swelling, due to effusion (fluid collection) in a synovial sac.
Time Frame: Baseline, Months 6, 12, 18, 30, 42, 54 and 66
Population: FAS included all recruited participants who were either initiated or were already receiving etanercept. The 'n' is signifying those participants who were evaluated for this measure at the specified time points.
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Etanercept
Number analyzed (Participants) | 25
joints
  Baseline | 26.5 (15.7)
  Change at Month 6 (n= 14) | -20.2 (15.8)
  Change at Month 12 (n= 15) | -20.3 (14.1)
  Change at Month 18 (n= 19) | -21.4 (15.2)
  Change at Month 30 (n= 22) | -19.5 (16.7)
  Change at Month 42 (n= 20) | -24.4 (16.3)
  Change at Month 54 (n= 18) | -24.3 (16.2)
  Change at Month 66 (n= 13) | -22.8 (19.2)

4. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire (HAQ) Score at Months 6, 12, 18, 30, 42, 54 and 66
Description: HAQ is a measure of functional limitations. Participants were rated on 4 point scale with scores as 'normal' (no difficulty = 0), 'adequate' (some difficulty = 1), 'limited' (much difficulty = 2), and 'unable to do' (= 3) based on degree of difficulty they experienced with 20 tasks grouped into 8 areas of dressing, rising, hygiene, reach, walking, eating, grip and activities. HAQ total possible score ranged from 0 (no difficulty) to 60 (unable to do).
Time Frame: Baseline, Months 6, 12, 18, 30, 42, 54 and 66
Population: FAS included all recruited participants who were either initiated or were already receiving etanercept. 'N' (number of participants analyzed) is signifying those participants who were evaluable for this measure. The 'n' is signifying those participants who were evaluated for this measure at the specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 18
units on a scale
  Baseline | 32.4 (12.0)
  Change at Month 6 (n= 6) | -13.7 (8.4)
  Change at Month 12 (n= 9) | -17.0 (7.5)
  Change at Month 18 (n= 10) | -17.8 (9.8)
  Change at Month 30 (n= 11) | -10.4 (14.5)
  Change at Month 42 (n= 9) | -20.0 (15.3)
  Change at Month 54 (n= 8) | -16.6 (14.3)
  Change at Month 66 (n= 2) | -26.5 (13.4)

5. Secondary Outcome: Mean Dose of Concomitant Methotrexate (MTX) and Steroids
Time Frame: Baseline up to Month 66
Population: Data was not analyzed due to low number of participants.
Measure: Mean (Standard Deviation); unit: milligram (mg)
Arm/Group | Etanercept
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Etanercept
Serious Adverse Events (participants affected / at risk) | 6/25
Other Adverse Events (participants affected / at risk) | 13/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=25)
Angioneurotic oedema (General disorders) | 1
Myocardial infarction (General disorders) | 1
Leucopenia (General disorders) | 1
Neutropenia (General disorders) | 1
Liver function test abnormal (General disorders) | 1
Knee arthroplasty (General disorders) | 1
Breast cancer (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=25)
Allergy (General disorders) | 1
Fatigue (General disorders) | 5
General discomfort with hypotension (General disorders) | 1
Injection site reaction (General disorders) | 2
Sleep Trouble (General disorders) | 1
Vertigo (General disorders) | 1
Fracture left clavicle (General disorders) | 1
Osteoporosis fractures (General disorders) | 1
Synoviorthesis knee (General disorders) | 1
High blood pressure (General disorders) | 1
Constipation (General disorders) | 2
Diarrhea (General disorders) | 2
Flatulence (General disorders) | 1
Increased hepatic enzymes (General disorders) | 1
Rectorragies (General disorders) | 1
Increased intra-ocular pressure (General disorders) | 1
Ocular dryness (General disorders) | 1
Aphtosis (General disorders) | 1
Buccal dryness (General disorders) | 1
Hypersensitivity tooth (General disorders) | 1
Bronchopneumopathy recurrent (General disorders) | 1
Dyspnea (General disorders) | 1
Pulmonary oedema (General disorders) | 1
Laryngitis (General disorders) | 1
Sinusitis (General disorders) | 1
Pruritus (General disorders) | 1
Nose and skin bleeding (General disorders) | 1
Zona (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.